CLINICAL TRIAL: NCT02531763
Title: Behavioral Economics Framingham Incentive Trial: A Randomized Controlled Trial
Brief Title: Behavioral Economics Framingham Incentive Trial (BE FIT)
Acronym: BEFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Boston University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1ZIAHL006094-05 (NIH); HHSN268201500056P (Other: NHLBI)
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Physical Activity
Keywords: mHealth; behavioral economics; social incentives
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): FHS participants who enrolled with family member will not receive the social incentive intervention and will participate individually but will set a daily step goal and receive daily feedback on whether he or she achieved the goal or not.
- Intervention (Active Comparator): FHS participants who enrolled with a family member will be placed on a team as connected individuals (both in the same family) who will set a daily step goal, receive daily feedback on whether they achieved their goal, and receive the social incentive intervention.
  Interventions: Behavioral: Social incentive intervention

INTERVENTIONS:
Behavioral: Social incentive intervention — Participant sign a pre-commitment pledge to try to achieve their goal. They are entered into a game with their teammate in which they have the chance to earn points and advance through levels (bronze, silver, gold, platinum). At the end, those in gold or platinum will receive a coffee mug as a reward
  Arms: Intervention

SUMMARY:
BE FIT (Behavioral Economics Framingham Incentive Trial) is a pilot study to test the deployment of a social incentive intervention using the Framingham Heart Study (FHS) Offspring, Generation 3, and Omni cohorts to increase physical activity (PA). The investigators will leverage the strength of FHS by recruiting trios and nuclear families to test whether social connectedness increases PA. The investigators will utilize a randomized controlled trial design. The investigators will test a social incentive intervention strategy using a team-based design in which participants work together to jointly achieve their PA goals, and a social connectedness intervention.

DETAILED DESCRIPTION:
Physical inactivity is associated with cardiovascular disease (CVD) risk factors, including obesity, diabetes, dyslipidemia, and hypertension, and an increased risk for CVD and death. In the Framingham Heart Study (FHS) Third Generation (Gen 3) and multiethnic Omni 2 cohort participants, objectively measured accelerometry physical activity (PA) data showed that moderate to vigorous PA was associated with healthier CVD risk factor profiles.6 Despite the health benefits of engaging in PA, only about half of FHS participants are achieving U.S. recommended aerobic PA guidelines, consistent with the low rates observed in adults nationally. Experts estimate that increasing PA by only 10% would annually save ½ million lives worldwide.

There has been a lot of interest in using "social" or team-based designs to increase PA. Prior evaluations of the FHS found that rates of smoking and obesity were associated with social connectedness within social networks. Evidence from other industries has found that interventions using social comparisons feedback to change electricity use were effective, but only if paired with appropriate social approval or disapproval. PA interventions could leverage such social incentives to design interventions that increase peer support, accountability, and unity towards a common goal. In five pilot studies conducted in 2014 at the University of Pennsylvania, the investigators have found that different incentive and feedback designs resulted in differential effectiveness. These preliminary data support the notion that careful testing of alternative social incentive combinations are important to conduct before deciding which intervention to scale more broadly.

The rapidly expanding availability of mobile technologies provides a resource effective way to implement social incentive interventions to improve health. Many types of health devices (e.g. glucometers, pedometers) provide individual feedback on performance (e.g. blood sugar or step count). With wireless devices it is technologically feasible to provide relative feedback at periodic intervals. However, utilizing mobile health (mHealth) devices is rarely done and could represent a significant opportunity to improve health behavior at low cost. For our study, the investigators will leverage the University of Pennsylvania's NIH-funded Way to Health infrastructure. The platform incorporates automated inputs from wireless devices to capture behavior and deliver automated feedback to participants. While conducting the 5 pilot studies noted above, the investigators found that most smartphones and wearable devices were accurate for tracking physical activity data.

The investigators are conducting a pilot study and leveraging information acquired through our Digital Connectedness Survey to test the deployment of a social incentive intervention using the FHS Offspring, Generation 3, and Omni cohorts to increase PA. The investigators will leverage the strength of FHS by recruiting trios and nuclear families to test whether social connectedness increases PA. The investigators will utilize a randomized controlled trial design. The investigators will test a social incentive intervention strategy using a team-based design in which participants work together to jointly achieve their PA goals, and a social connectedness intervention. The primary outcome of the intervention pilot study will be the proportion of individual participant-days that the goal is achieved over a 12-week intervention period. Individuals find PA maintenance challenging and PA sustainability has not been studied systematically. As a secondary aim of the intervention study, the investigators will examine PA goal achievement durability for 12 weeks after the intervention ends.

Specific Aims:

Aim 1. To test the feasibility of using a team-based social incentive intervention to increase PA in FHS participants. H1: The demographic and clinical characteristics of individuals who agrees to be randomized are younger and healthier than those who do not agree to participate. H2: FHS participants who elect the Fitbit in place of the Moves app will differ based on demographic and clinical characteristics.

Aim 2. To evaluate the effectiveness of a team-based social incentive intervention to achieve PA goals among connected individuals on a team compared to a control group of individuals. H4: A team-based social incentive intervention comprised of connected individuals on a team is more effective for achieving PA goals than a control group of individuals.

Secondary Aim. To evaluate whether differences in achieving PA goals between study arms during the 12-week intervention are sustained during the 12-week follow-up period. H6: PA levels in the 12-week follow-up will decline for all arms but remain different in a similar fashion to that during the intervention period.

This study has the potential to address the major public health problem of sedentary lifestyle, with its consequent increased risks of obesity and CVD risk factor progression. The investigators bring together a multi-disciplinary team with expertise in PA, CVD epidemiology, biostatistics, and behavioral economics. The investigators propose an innovative linking of a classical randomized clinical trial (RCT) design with the many strengths of the epidemiological FHS. This pilot RCT will examine the effectiveness of different approaches to leveraging social incentives to improve health behaviors, an area with considerable promise for increasing the effectiveness of a variety of health interventions. Ultimately the goal is to leverage this pilot study to implement a larger study in the FHS. The investigators also anticipate ultimately linking these results with the extant FHS genetics databases.

ELIGIBILITY:
Inclusion Criteria:

1. FHS study members from any of the existing cohorts (Offspring, Gen 3, Omni groups 1)
2. Must have active email address
3. Must have participated in the FHS Digital Connectedness Survey
4. Must have at least 2 family members in the FHS

Exclusion Criteria:

1. Not currently participating in any other physical activity studies.
2. Not told by a physician not to exercise.
3. Not currently pregnant.
4. Not had at least one fall with significant injury in the past year.
5. Not had any surgical procedures in the participants' legs that would prohibit physical activity.
6. Not have any other medical conditions or other reasons to prevent participation in a 6 month physical activity program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
proportion of days achieving their step goals over intervention period. | 12 weeks

SECONDARY OUTCOMES:
Mean daily steps adjusted for baseline step count | Weeks 1 to 12, and weeks 13 to 24
Proportion participant-days achieving step goals | Weeks 13 to 24

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Fox, MD MPH, Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)

REFERENCES:
- [Derived] Patel MS, Benjamin EJ, Volpp KG, Fox CS, Small DS, Massaro JM, Lee JJ, Hilbert V, Valentino M, Taylor DH, Manders ES, Mutalik K, Zhu J, Wang W, Murabito JM. Effect of a Game-Based Intervention Designed to Enhance Social Incentives to Increase Physical Activity Among Families: The BE FIT Randomized Clinical Trial. JAMA Intern Med. 2017 Nov 1;177(11):1586-1593. doi: 10.1001/jamainternmed.2017.3458. PMID 28973115